CLINICAL TRIAL: NCT04785027
Title: Comparison of PSORI-CM01 Formula vs Gu Ben Hua Yu Formula Combined With Expanded Allogeneic Adipose-derived Mesenchymal Stem Cells in Patients With Moderate to Severe Psoriasis: a Pilot Study for a Randomized Controlled Trial
Brief Title: Comparison of PSORI-CM01 Formula vs Gu Ben Hua Yu Formula Combined With AD-MSCs in Psoriasis
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangdong Provincial Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Chuanjian Lu, Professor, Guangdong Provincial Hospital of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S2020-01-01
Record Dates: First submitted 2021-02-28; First posted 2021-03-05 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Traditional Chinese Medicine; Drug Effect; Drug Safety; Psoriasis; Mesenchymal Stromal Cells
Keywords: Traditional Chinese Medicine; Mesenchymal Stem Cells; Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PSORI-CM01 group (Other): Expanded Allogeneic Adipose-derived multipotent mesenchymal stem cells(AD-MSCs) will be administered by intravenous drip at a dose of 2×10 ^ 6 cells/kg at week 0, week 2, week 4, week 6, week 8 with a total of 5 times.
  PSORI-CM01 formula will be orally administrated once a day for 12 weeks excpet the day for the infusion of AD-MSCs.
  Interventions: Drug: PSORI-CM01 formula; Biological: adipose-derived multipotent mesenchymal stem cells
- Gu Ben Hua Yu group (Experimental): Expanded Allogeneic Adipose-derived multipotent mesenchymal stem cells(AD-MSCs) will be administered by intravenous drip at a dose of 2×10 ^ 6 cells/kg at week 0, week 2, week 4, week 6, week 8 with a total of 5 times.
  Gu Ben Hua Yu formula will be orally administrated once a day for 12 weeks excpet the day for the infusion of AD-MSCs.
  Interventions: Drug: Gu Ben Hua Yu formula; Biological: adipose-derived multipotent mesenchymal stem cells

INTERVENTIONS:
Drug: PSORI-CM01 formula — PSORI-CM01 formula will be orally administrated once a day for 12 weeks excpet the day for the infusion of AD-MSCs
  Other Names: Chinese Herbal Medicine
  Arms: PSORI-CM01 group
Drug: Gu Ben Hua Yu formula — Gu Ben Hua Yu formula will be orally administrated once a day for 12 weeks excpet the day for the infusion of AD-MSCs
  Other Names: Chinese Herbal Medicine
  Arms: Gu Ben Hua Yu group
Biological: adipose-derived multipotent mesenchymal stem cells — AD-MSCs (adipose-derived multipotent mesenchymal stem cells) will be infused intravenously at a dose of 2 million cells/kg
  Other Names: stem cells; AD-MSCs

SUMMARY:
The purpose of this study is to evaluate and compare the safety and efficacy of PSORI-CM01 formula vs Gu Ben Hua Yu formula combined with Expanded Allogeneic AD-MSCs in patients with moderate to severe psoriasis. And it explores the expectations of patients for the treatment of traditional Chinese medicine combined with stem cells and their expectations to participate in this study. The trial would provide preliminary data for large sample clinical randomized controlled trials.

DETAILED DESCRIPTION:
Psoriasis is an immune-mediated, genetic disease manifesting in the skin or joints or both. Treatment modalities are chosen on the basis of disease severity, relevant comorbidities, patient preference. For moderate to severe psoriasis, phototherapy, systemic therapy and biologic immune modifying agents are recommended, but all of them have some drawbacks or limitations. Until now, no curative treatment is available. Therefore, it is important to find new treatment for psoriasis.

As current experience and cases of AD-MSCs in the treatment of psoriasis are still relatively small, and it is unknown about their safety and efficacy combined with traditional medicine in the treatment of psoriasis.

This study designed a randomized controlled trial to compare PSORI-CM01 formula vs Guben Huayu formula combined with expanded allogeneic adipose-derived mesenchymal stem cells in the treatment of psoriasis. The purpose of this study is to evaluate and compare the safety and efficacy of PSORI-CM01 formula vs Gu Ben Hua Yu formula combined with Expanded Allogeneic AD-MSCs in patients with moderate to severe psoriasis. And it also aims to determine the feasibility and the potential of the protocol for the full-scale randomized controlled trial (RCT).

Therefore, 16 subjects will be enrolled in this study and their expectations for the treatment of traditional Chinese medicine combined with stem cells and their experience to participate in this study will be interviewed.

ELIGIBILITY:
Inclusion Criteria:

1.patients with psoriasis vulgaris(PASI > 7 or BSA >10%); 2.18 to 65 years old; 3.written/signed informed consent.

Exclusion Criteria:

1. The skin lesions are seen alone on the patient's face, scalp, nails, wrinkles, glans, mucous membranes, palmar and plantar or guttate psoriasis;
2. Acute progressive psoriasis, and erythroderma tendency;
3. current (or within 1 year) pregnancy or lactation;
4. current significant anxiety or depression with the Self-rating Anxiety Scale (SAS) > 50 or the Self-rating Depression Scale (SDS) > 53, or with other psychiatric disorders;
5. With history of primary cardiovascular, respiratory, digestive, urinary, endocrinologic and hematologic diseases, which can't be controlled through ordinary treatments. Those who with malignant diseases,infections, electrolyte imbalance, acid-base disturbance. Patients with clinical test results listed below: abnormal serum calcium level ( Ca2+> 2.9 mmol/L or < 2 mmol/L);AST or ALT 2 times more than normal upper limit; Creatinine and cystatin C more than normal upper limit;Hemoglobin elevates 20g/L more than normal upper limit,or hemoglobin reduction to anemia; Platelet count less than 75.0*10^9/L; White blood cell less than 3.0*10^9/L; Or any other abnormal laboratory test results, assessed by investigators, that are not suitable for this clinical study;
6. Patients with malignant tumors, or when they were enrolled with abnormal tumor markers or with other organ dysfunction;
7. allergy to anything else ever before;
8. current registration in other clinical trials or participation within a month;
9. topical treatments (i.e. corticosteroids or retinoic acid or Vitamin D analogs ) within 2 weeks; systemic therapy or phototherapy (ultraviolet radiation B,UVB) and psoralen combined with ultraviolet A (PUVA) within 4 weeks; biological therapy within 12 weeks;
10. medical conditions assessed by investigators, that are not suitable for this clinical study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2021-03-17 (Actual); Primary Completion 2021-06-17 (Actual); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
PASI score improvement rate | 12 weeks (plus or minus 3 days) after treatment.
  PASI score improvement rate = (PASI score before intervention - PASI score after intervention)/PASI score before intervention ×100% PASI scores the average redness, thickness, and scaliness of the lesions (0-4 scale), weighted by the area of involvement. PASI scores range from 0 to 72. The higher the score, the worse the disease.

SECONDARY OUTCOMES:
PASI (Psoriasis Area and Severity Index) | 12 weeks (plus or minus 3 days) after treatment.
  The improvement in PASI score from baseline after treatment. PASI scores the average redness, thickness, and scaliness of the lesions (0-4 scale), weighted by the area of involvement. PASI scores range from 0 to 72. The higher the score, the worse the disease.
Relapse rate in treatment period / follow-up period | 12 weeks (plus or minus 3 days) after treatment.
  Relapse can be defined only for patients who achieve PASI-50，and occurs when the improvement in the PASI score falls below 50 percent from the baseline PASI score.
PASI-50 | 12 weeks (plus or minus 3 days) after treatment.
  The proportion of patients who achieve at least 50 percent improvement in PASI score from baseline.
PASI-75 | 12 weeks (plus or minus 3 days) after treatment.
  The proportion of patients who achieve at least 75 percent improvement in PASI score from baseline.
Pruritus Scores on the Visual Analogue Scale | 12 weeks (plus or minus 3 days) after treatment.
  Pruritus was assessed using the Visual Analogue Scales; The Scale scores ranged from 0-10. The higer the scores were, the more itching the patient suffered.
BSA | 12 weeks (plus or minus 3 days) after treatment.
  the Body Surface Area
DLQI (Dermatology Life Quality Index) | 12 weeks (plus or minus 3 days) after treatment.
  the score of Dermatology Life Quality Index. Dermatology Life Quality Index (DLQI) is a self-administered 10-item questionnaire. It covers Symptoms and feelings, Daily activities, Leisure, Work and school, Personal relationships, and Treatment. The higher the score, the worse the quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Chuanjian Lu, PhD, Principal Investigator — Guangdong Provincial Hospital of Traditional Chinese Medicine
Locations (1):
- Guangdong Provincial Hospital of Traditional Chinese Medicine, Guangzhou, Guangdong, China